CLINICAL TRIAL: NCT02722499
Title: Financial Incentives Augmented Telephone Education and Skills Trial in African Americans With Diabetes (FITEST)
Brief Title: Financial Incentives Telephone Education and Skills Trial in African Americans With Diabetes (FITEST)
Acronym: FITEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Leonard Ehianu Egede, Professor & Chair, Department of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00021791
Record Dates: First submitted 2016-03-23; First posted 2016-03-30 (Estimated); Results first posted 2021-11-05 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus; Type 2 Diabetes Mellitus; Adult-Onset Diabetes Mellitus; Non-Insulin-Dependent Diabetes Mellitus; Noninsulin Dependent Diabetes Mellitus, Type II
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset; Diabetes Mellitus, Non-Insulin-Dependent; Diabetes Mellitus, Noninsulin Dependent; Diabetes Mellitus, Type II; African American; Blacks; non-Hispanic Blacks; Randomized Control Trial; Controlled Clinical Trial; Behavioral Research; Behavioral Medicine
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Frequency Financial Incentive (Experimental): This arm will receive telephone delivered diabetes education and skills training in combination with the high frequency incentive structure
  Interventions: Behavioral: High Frequency Financial Incentive
- Moderate Frequency Financial Incentive (Experimental): This arm will receive telephone delivered diabetes education and skills training in combination with the moderate frequency incentive structure
  Interventions: Behavioral: Moderate Frequency Financial Incentive
- Low Frequency Financial Incentive (Experimental): This arm will receive telephone delivered diabetes education and skills training in combination with the low frequency incentive structure
  Interventions: Behavioral: Low Frequency Financial Incentive

INTERVENTIONS:
Behavioral: High Frequency Financial Incentive — 1. Diabetes Education/Skills Component. Subjects will receive weekly telephone-delivered diabetes/skills training for 12 weeks with home telemonitoring.
  2. High Frequency Financial Incentive: the high frequency incentive structure will receive a reward for uploading glucose measurements, attending educational sessions, and absolute percentage drops in HbA1c from baseline at 3-month follow-up, up to $300. Each week participants can receive up to $10 for uploading glucose measurements and having good glucose control throughout the week. If they upload measurements every day of the week and their average glucose measurements at the end of the week are 150 or below they will receive an additional $3. Participants can also earn $5 each week if they attend the educational session. After 3 months, if their HbA1c has dropped 2% from baseline, or absolute HbA1c is 7%, they will receive a reward of $130, for a 1% drop, or an absolute HbA1c between 7 and 8 they will receive a reward of $65.
  Other Names: Group 3
  Arms: High Frequency Financial Incentive
Behavioral: Moderate Frequency Financial Incentive — 1. Diabetes Education/Skills Component. Subjects will receive weekly telephone-delivered diabetes/skills training for 12 weeks with home telemonitoring.
  2. Moderate Frequency Financial: the moderate frequency incentive structure will receive a reward for uploading glucose measurements, and absolute percentage drops in HbA1c from baseline at 3-month follow-up, up to $300. Each week participants can receive up to $10 for uploading glucose measurements and having good glucose control throughout the week. For each day they upload at least one glucose measurement, they will receive $1 (up to $7 at the end of the week). If they upload measurements every day of the week and their average glucose measurements at the end of the week are 150 or below they will receive an additional $3. After 3 months, if their HbA1c has dropped 2% from baseline, or absolute HbA1c is 7%, they will receive a reward of $170, for a 1% drop, or an absolute HbA1c between 7 and 8 they will receive a reward of $85
  Other Names: Group 2
  Arms: Moderate Frequency Financial Incentive
Behavioral: Low Frequency Financial Incentive — 1. Diabetes Education/Skills Component. Subjects will receive weekly telephone-delivered diabetes/skills training for 12 weeks with home telemonitoring.
  2. Low Frequency Financial Incentive: the low frequency incentive structure will receive a reward for absolute percentage drops in HbA1c from baseline at 3-month follow-up, up to $300. After 3 months, if their HbA1c has dropped 2% from baseline, or absolute HbA1c is 7%, they will receive a reward of $300, for a 1% drop, or an absolute HbA1c between 7 and 8 they will receive a reward of $150.
  Other Names: Group 1
  Arms: Low Frequency Financial Incentive

SUMMARY:
The aim of this study is to test the efficacy of financial incentives augmented telephone-delivered diabetes education and skills training intervention in improving HbA1c levels in African Americans (AA) with type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
African Americans with T2DM have higher prevalence of diabetes, poorer metabolic control, and greater risk for complications and death compared to White Americans. HbA1c is the primary marker for glycemic control and is a strong independent predictor of development of complications and increased mortality in T2DM. Key self-care behaviors that influence glycemic control (and HbA1c) include diet, physical activity, self-monitoring of blood glucose and medication adherence. Systematic review of multiple RCTs show that self-care interventions that include diabetes education and skills training are effective in improving metabolic control in diabetes. Recent findings indicate that patients with diabetes, especially ethnic minority patients, prefer telephone-delivered diabetes education to group visits or internet-based education. Multiple RCTs have documented the effectiveness of telephone-delivered self-care interventions in T2DM.

The overarching aim of this proposal is test the efficacy of three financial incentive structures in combination with technology intensified diabetes education and skills training intervention on blood pressure and quality of life in AAs with T2DM. 60 AAs with T2DM will be randomized to three groups with varying frequency of financial incentives: 1) High Frequency: financial incentives for weekly uploads plus average glucose, incentives for weekly attendance to educational sessions, and incentives at the end of the study for meeting HbA1c goals 2) Moderate Frequency: financial incentives for weekly uploads plus average glucose, and incentives at the end of the study for meeting HbA1c goals, and 3) Low Frequency: financial incentives at the end of the study for meeting HbA1c goals.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years
* Clinical diagnosis of T2DM and HbA1c ≥8% at the screening visit
* Self-identified as AA
* Subject must be willing to use the FORA monitoring system for 3 months
* Subjects must be able to communicate in English
* Subjects must have access to a telephone (landline for data uploads) for the study period

Exclusion Criteria:

* Mental confusion on interview suggesting significant dementia
* Participation in other diabetes clinical trials
* Alcohol or drug abuse/dependency
* Active psychosis or acute mental disorder
* Life expectancy <12 months

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E Egede, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Result] Egede LE, Campbell JA, Walker RJ, Dawson AZ, Williams JS. Financial incentives to improve glycemic control in African American adults with type 2 diabetes: a pilot randomized controlled trial. BMC Health Serv Res. 2021 Jan 13;21(1):57. doi: 10.1186/s12913-020-06029-0. PMID 33435969
- [Result] Egede LE, Walker RJ, Dismuke-Greer CE, Pyzyk S, Dawson AZ, Williams JS, Campbell JA. Cost-effectiveness of financial incentives to improve glycemic control in adults with diabetes: A pilot randomized controlled trial. PLoS One. 2021 Mar 18;16(3):e0248762. doi: 10.1371/journal.pone.0248762. eCollection 2021. PMID 33735275

RESULTS

PARTICIPANT FLOW:
Groups:
- High Frequency Financial Incentive: This arm will receive telephone delivered diabetes education and skills training in combination with the high frequency incentive structure
  High Frequency Financial Incentive: 1. Diabetes Education/Skills Component. Subjects will receive weekly telephone-delivered diabetes/skills training for 12 weeks with home telemonitoring.
  2. High Frequency Financial Incentive: the high frequency incentive structure will receive a reward for uploading glucose measurements, attending educational sessions, and absolute percentage drops in HbA1c from baseline at 3-month follow-up, up to $300. Each week participants can receive up to $10 for uploading glucose measurements and having good glucose control throughout the week. If they upload measurements every day of the week and their average glucose measurements at the end of the week are 150 or below they will receive an additional $3. Participants can also earn $5 each week if they attend the educational session. After 3 months, if their HbA1c has dropped 2% from baseline, or absolute HbA1c is 7%, they will receive a reward of $130, for a 1% drop, or an absolute HbA1c between 7 and 8 they will receive a reward of $65.
- Moderate Frequency Financial Incentive: This arm will receive telephone delivered diabetes education and skills training in combination with the moderate frequency incentive structure
  Moderate Frequency Financial Incentive: 1. Diabetes Education/Skills Component. Subjects will receive weekly telephone-delivered diabetes/skills training for 12 weeks with home telemonitoring.
  2. Moderate Frequency Financial: the moderate frequency incentive structure will receive a reward for uploading glucose measurements, and absolute percentage drops in HbA1c from baseline at 3-month follow-up, up to $300. Each week participants can receive up to $10 for uploading glucose measurements and having good glucose control throughout the week. For each day they upload at least one glucose measurement, they will receive $1 (up to $7 at the end of the week). If they upload measurements every day of the week and their average glucose measurements at the end of the week are 150 or below they will receive an additional $3. After 3 months, if their HbA1c has dropped 2% from baseline, or absolute HbA1c is 7%, they will receive a reward of $170, for a 1% drop, or an absolute HbA1c between 7 and 8 they will receive a reward of $85
- Low Frequency Financial Incentive: This arm will receive telephone delivered diabetes education and skills training in combination with the low frequency incentive structure
  Low Frequency Financial Incentive: 1. Diabetes Education/Skills Component. Subjects will receive weekly telephone-delivered diabetes/skills training for 12 weeks with home telemonitoring.
  2. Low Frequency Financial Incentive: the low frequency incentive structure will receive a reward for absolute percentage drops in HbA1c from baseline at 3-month follow-up, up to $300. After 3 months, if their HbA1c has dropped 2% from baseline, or absolute HbA1c is 7%, they will receive a reward of $300, for a 1% drop, or an absolute HbA1c between 7 and 8 they will receive a reward of $150.
Period: Overall Study
Arm/Group | High Frequency Financial Incentive | Moderate Frequency Financial Incentive | Low Frequency Financial Incentive
Started | 20 | 20 | 20
Completed | 18 | 20 | 19
Not Completed | 2 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Frequency Financial Incentive | Moderate Frequency Financial Incentive | Low Frequency Financial Incentive | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.6) | 57.4 (8.8) | 58.1 (14.1) | 57.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 15 | 39
  Male | 8 | 8 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 20 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 20 | 20 | 20 | 60
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 10.4 (2.3) | 9.9 (1.3) | 10.1 (2.1) | 10.1 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: Hemoglobin A1c (HbA1c): blood specimens will be collected at the screening visit, as well as the 3-months. Time points used in calculation are baseline to 3 month.
Time Frame: Baseline to 3 months
Population: 20 subjects randomized to each arm, but 18 included in final analysis in high frequency, 20 in moderate frequency and 19 in low frequency arms respectively
Measure: Mean (95% Confidence Interval); unit: mean change from baseline
Arm/Group | High Frequency Financial Incentive | Moderate Frequency Financial Incentive | Low Frequency Financial Incentive
Number analyzed (Participants) | 18 | 20 | 19
mean change from baseline | -1.73 [-2.55 to -0.92] | -1.73 [-2.48 to -0.99] | -1.25 [-1.98 to -0.52]

2. Secondary Outcome: Resource Utilization and Cost
Description: Resource Utilization & Cost: Information on hospitalizations, physician/professional visits, and medications will be captured. Time points used in calculation are baseline to 3 month.
Time Frame: Baseline to 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | High Frequency Financial Incentive | Moderate Frequency Financial Incentive | Low Frequency Financial Incentive
Number analyzed (Participants) | 18 | 20 | 19
US Dollars | 3315.45 (2014.43) | 4649.68 (5393.52) | 3765.57 (2765.57)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | High Frequency Financial Incentive | Moderate Frequency Financial Incentive | Low Frequency Financial Incentive
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT02722499/Prot_SAP_000.pdf